CLINICAL TRIAL: NCT00001040
Title: Double-Blind, Randomized, Phase II Study of Ro 31-8959 Plus Zidovudine (AZT) Versus AZT Plus Zalcitabine (Dideoxycytidine; ddC) Versus Ro 31-8959 Plus AZT Plus ddC
Brief Title: Comparison of Ro 31-8959 Plus Zidovudine (AZT) Versus AZT Plus Zalcitabine (ddC) Versus Ro 31-8959 Plus AZT Plus ddC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 229; NV14255D; FDA 123A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Saquinavir; HIV Protease Inhibitors
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Saquinavir; Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Saquinavir
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
PRIMARY: To determine the efficacy and toxicity of three treatment regimens: saquinavir mesylate (Ro 31-8959) plus zidovudine (AZT) vs. AZT plus zalcitabine (dideoxycytidine; ddC) vs. Ro 31-8959 plus AZT plus ddC.

SECONDARY: To investigate the pharmacokinetics and effects on various clinical parameters of the three regimens.

ELIGIBILITY:
Inclusion Criteria

Prior Medication: Required:

* At least 4 months total of AZT at some point in the past, alone or in combination with other antiretroviral therapy.

Patients must have:

* HIV seropositivity.
* Diagnosis of AIDS, ARC, PGL, or asymptomatic infection.
* CD4 count > 50 to <= 300 cells/mm3.
* Life expectancy of at least 6 months.
* Prior AZT therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Acute serious opportunistic infections requiring immediate treatment, including (but not limited to) tuberculosis, CMV, cryptococcal meningitis, disseminated MAC, cerebral toxoplasmosis, and Pneumocystis carinii pneumonia.
* Known intolerance to Ro 31-8959, AZT, or ddC.
* Symptoms suggestive of pancreatitis.
* Moderate or severe peripheral neuropathy as evidenced by discomfort from numbness, tingling, burning or pain of the extremities or any related symptoms that are accompanied by an objective finding.
* Visceral Kaposi's sarcoma.
* Lymphoma that will require therapy within the next 6 months.
* Transfusion dependence.

Concurrent Medication:

Excluded:

* Investigational or antineoplastic agents.

Concurrent Treatment:

Excluded:

* Radiotherapy (other than local skin radiotherapy).
* Transfusions.

Prior Medication:

Excluded:

* Any antiretroviral agent (other than AZT) or immunomodulatory therapy within 14 days prior to study entry.
* Prior treatment with an HIV proteinase inhibitor.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Primary Completion 1994-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Collier AC, Study Chair; Corey L, Study Chair
Locations (10):
- United States (10):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Northwestern Univ Med School, Chicago, Illinois
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Ohio State Univ Hosp, Columbus, Ohio
  - Girard Med Ctr, Philadelphia, Pennsylvania
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Schapiro JM, Lawrence J, Speck R, Winters MA, Efron B, Coombs RW, Collier AC, Merigan TC. Resistance mutations to zidovudine and saquinavir in patients receiving zidovudine plus saquinavir or zidovudine and zalcitabine plus saquinavir in AIDS clinical trials group 229. J Infect Dis. 1999 Jan;179(1):249-53. doi: 10.1086/314541. PMID 9841849
- [Background] Brambilla D, Coombs R, Bremer JW, Reichelderfer PS, Kalish L, Shapiro DE. The contributions of assay variation and biological variation to the variability of HIV RNA measurements in serially collected clinical specimens. Int Conf AIDS. 1998;12:805 (abstract no 42163)
- [Background] Collier AC, Coombs RW, Schoenfeld DA, Bassett R, Baruch A, Corey L. Combination therapy with zidovudine, didanosine and saquinavir. Antiviral Res. 1996 Jan;29(1):99. doi: 10.1016/0166-3542(95)00928-0. PMID 8721557
- [Background] Collier AC, Coombs RW, Timpone J, Schoenfeld DA, Bassett R, Baruch A, Corey L. Comparative study of Ro 31-8959 and zidovudine (ZDV) vs. ZDV and zalcitabine (ddC) vs. Ro 31-8959, ZDV, and ddC. The ACTG 229 Protocol Team. Int Conf AIDS. 1994 Aug 7-12;10(1):21 (abstract no 058B)
- [Background] Noble S, Faulds D. Saquinavir. A review of its pharmacology and clinical potential in the management of HIV infection. Drugs. 1996 Jul;52(1):93-112. doi: 10.2165/00003495-199652010-00007. PMID 8799687
- [Background] Vanhove GF, Gries JM, Verotta D, Sheiner LB, Coombs R, Collier AC, Blaschke TF. Exposure-response relationships for saquinavir, zidovudine, and zalcitabine in combination therapy. Antimicrob Agents Chemother. 1997 Nov;41(11):2433-8. doi: 10.1128/AAC.41.11.2433. PMID 9371346
- [Background] Collier AC, Coombs RW, Schoenfeld DA, Bassett RL, Timpone J, Baruch A, Jones M, Facey K, Whitacre C, McAuliffe VJ, Friedman HM, Merigan TC, Reichman RC, Hooper C, Corey L. Treatment of human immunodeficiency virus infection with saquinavir, zidovudine, and zalcitabine. AIDS Clinical Trials Group. N Engl J Med. 1996 Apr 18;334(16):1011-7. doi: 10.1056/NEJM199604183341602. PMID 8598838
- [Background] Fischl MA, Stanley K, Collier AC, Arduino JM, Stein DS, Feinberg JE, Allan JD, Goldsmith JC, Powderly WG. Combination and monotherapy with zidovudine and zalcitabine in patients with advanced HIV disease. The NIAID AIDS Clinical Trials Group. Ann Intern Med. 1995 Jan 1;122(1):24-32. doi: 10.7326/0003-4819-122-1-199501010-00004. PMID 7985892
- [Background] Schapiro JM, Lawrence J, Speck R, Winters MA, Coombs R, Collier AC, Efron B, Merigan TC. HIV RNA and resistance mutations to saquinavir and zidovudine in patients receiving dual versus triple combination therapy. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:154 (abstract no 401)